CLINICAL TRIAL: NCT00517231
Title: Cytokines and Acute Phase Reactants as Markers of Pulmonary Tuberculosis Treatment
Status: Withdrawn | Type: Observational
Why Stopped: The investigator left the research center and the study was not carried out
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Other Study IDs: upeclin/HC/FMB-Unesp-pre02
Record Dates: First submitted 2007-08-14; First posted 2007-08-16 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Pulmonary Tuberculosis
Keywords: Pulmonary tuberculosis; Mycobacterium tuberculosis; Cytokines; Acute Phase Response; Treatment
MeSH Terms: conditions — Tuberculosis, Pulmonary; Acute-Phase Reaction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Tuberculosis is a highly prevalent chronic infectious disease caused by Mycobacterium tuberculosis. Cytokines are important biological mediators that regulate immune and inflammatory responses against the bacilli, witch include the acute phase response. Besides this, it becomes essential to determine markers of healing lesions, once this is currently carried out based on the clinical, radiological, and negative bacterioscopy.

DETAILED DESCRIPTION:
Tuberculosis is a highly prevalent chronic infectious disease caused by Mycobacterium tuberculosis. Cytokines are important biological mediators that regulate immune and inflammatory responses against the bacilli, witch include the acute phase response. Besides this, it becomes essential to determine markers of healing lesions, once this is currently carried out based on the clinical, radiological, and negative bacterioscopy. The propose of this work was to evaluate the production of IFN- γ in cell supernatants of peripheral blood mononuclear cells (PBMC) culture, TNF-α, IL-10 and TGF-b in cell supernatants of monocytes (MO) culture and biochemical (total proteins, albumin, globulin, α-1-acid glycoprotein and C-reactive protein) and hematological (VHS) serum parameters before and after 3 and 6 months of therapy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Mycobacterium tuberculosis infection

Exclusion Criteria:

* all other granulomatous or neoplastic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jussara Marcondes-Machado, PHD, Principal Investigator — Botucatu School of Medicine - Unesp